CLINICAL TRIAL: NCT03134313
Title: Accuracy of Noninvasive Rainbow Adhesive R1 Pulse Oximeter Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR18670-1029
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- R1-25 Sensor (Experimental): All subjects will be enrolled in the test group and will receive Rainbow Adhesive Noninvasive R1 Pulse Oximeter Sensor
  Interventions: Device: Rainbow Adhesive Noninvasive R1 Pulse Oximeter Sensor

INTERVENTIONS:
Device: Rainbow Adhesive Noninvasive R1 Pulse Oximeter Sensor

SUMMARY:
In this study, the concentration of hemoglobin will be measured using a noninvasive pulse oximeter sensor and compared with the hemoglobin value from a blood sample of the volunteer. The accuracy of a noninvasive hemoglobin sensor(s) will be assessed by comparison to hemoglobin measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Healthy

Exclusion criteria:

* Do not understand the study and the risks involved
* Deemed ineligible by study test personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12-12 (Actual); Primary Completion 2009-06-19 (Actual); Study Completion 2009-06-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- R1-25 Sensor: All subjects will be enrolled in the test group and will receive Rainbow Adhesive Noninvasive R1 Pulse Oximeter Sensor
  Rainbow Adhesive Noninvasive R1 Pulse Oximeter Sensor
Period: Overall Study
Arm/Group | R1-25 Sensor
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | R1-25 Sensor
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of SpHb on R1-25 by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square (Arms) error value. In order to obtain the Arms value, the blood sample hemoglobin value is subtracted from the pulse oximeter hemoglobin value for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours per subject
Measure: Number; unit: g/dL
Arm/Group | R1-25 Sensor
Number analyzed (Participants) | 25
g/dL | 1.0

ADVERSE EVENTS:
Arm/Group | R1-25 Sensor
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less